CLINICAL TRIAL: NCT02628574
Title: A Phase 1 Study of TRX518 Monotherapy and TRX518 in Combination With Gemcitabine, Pembrolizumab, or Nivolumab in Adults With Advanced Solid Tumors
Brief Title: Phase 1 Open-label Study of TRX518 Monotherapy and TRX518 in Combination With Gemcitabine, Pembrolizumab, or Nivolumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRX518-003
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors
Keywords: Metastatic; Stage III or IV; recurrent; refractory; solid tumors
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence | interventions — Gemcitabine; pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- TRX518 monotherapy (Parts A and B) (Experimental): Subjects receive an assigned dose of TRX518 administered intravenously one time per week or one time per cycle on a 21-day cycle
  Interventions: Drug: TRX518 monotherapy
- TRX518 with gemcitabine (Part C) (Experimental): Subjects receive an assigned dose of TRX518 (dosed one time per cycle) intravenously administered in combination with gemcitabine (dosed two times per cycle) on a 21-day cycle
  Interventions: Drug: TRX518 with gemcitabine
- TRX518 with pembrolizumab (Part D (Experimental): Subjects receive an assigned dose of TRX518 (dosed one time per cycle) intravenously administered in combination with pembrolizumab (dosed one time per cycle) on a 21-day cycle
  Interventions: Drug: TRX518 with pembrolizumab
- TRX518 with nivolumab (Part E) (Experimental): Subjects receive an assigned dose of TRX518 (dosed two times per cycle) intravenously administered in combination with nivolumab (dosed two times per cycle) on a 28-day cycle
  Interventions: Drug: TRX518 with nivolumab

INTERVENTIONS:
Drug: TRX518 monotherapy — comparison of different (ascending) doses of TRX518 monotherapy
  Arms: TRX518 monotherapy (Parts A and B)
Drug: TRX518 with gemcitabine — comparison of different (ascending) doses of TRX518 in combination with gemcitabine
  Arms: TRX518 with gemcitabine (Part C)
Drug: TRX518 with pembrolizumab — comparison of different (ascending) doses of TRX518 in combination with pembrolizumab
  Arms: TRX518 with pembrolizumab (Part D
Drug: TRX518 with nivolumab — comparison of different (ascending) doses of TRX518 in combination with nivolumab
  Arms: TRX518 with nivolumab (Part E)

SUMMARY:
This study will be conducted in 5 parts (Parts A, B, C, D and E).

Monotherapy Treatment:

Subjects ≥18 years with advanced solid tumors will be enrolled in the study. Monotherapy dose escalation will be performed in Part A. Cycle 1 data from each cohort will be evaluated for safety and dose-limiting toxicities (DLTs) prior to dose escalation. Subjects will be assigned to a cohort in the order screening is completed. Dose will depend upon the cohort in which a patient is enrolled and cohorts will be dosed consecutively by ascending dose. Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been identified, an expanded cohort will be enrolled (Part B).

Combination Treatment:

Subjects ≥18 years with advanced solid tumors will be enrolled in the study. Subjects will receive TRX518 in combination with gemcitabine (Part C), pembrolizumab (Part D), or nivolumab (Part E). Dose escalation will be performed for each part (Part Cesc, Part Desc, Part Eesc) and Cycle 1 data from each cohort will be evaluated for safety and dose-limiting toxicities (DLTs) prior to dose escalation. Subjects will be assigned to a cohort in the order screening is completed. Dose will depend upon the cohort in which a patient is enrolled and cohorts will be dosed consecutively by ascending dose. Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been identified, an expanded cohort will be enrolled (Part Cexp, Part Dexp, Part Eexp).

ELIGIBILITY:
Inclusion Criteria:

* Advanced Solid Malignancies: Histologically documented metastatic or locally advanced, incurable solid malignancy (Parts A and B); histologically documented metastatic or locally advanced, incurable solid malignancy for which gemcitabine is clinically appropriate (e.g., non-small cell lung, breast, ovarian, pancreatic, and renal cancer); histologically documented metastatic or locally advanced, incurable solid malignancy for which pembrolizumab (Part D) or nivolumab (Part E) is approved. NOTE: Parts D and E only: Subject has either (1) received treatment with pembrolizumab or nivolumab for ≥4 months with a best response of stable disease and plans to continue treatment with either pembrolizumab or nivolumab in accordance with package insert; or (2) is not currently taking, but is eligible for treatment with, pembrolizumab or nivolumab in accordance with the approved indications for each as referenced in the package insert.
* Expected survival of at least 12 weeks after dosing.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Evidence of adequate organ function by standard laboratory tests.
* All female subjects of child bearing age must be either surgically sterile, postmenopausal for at least 1 year, or using an acceptable method of contraception. Adequate contraception for both male and female subjects must be used from the beginning of the screening period until at least 8 weeks after the last dose of study drug.

Exclusion Criteria:

* Hematologic malignancies or multiple myeloma.
* Known, clinically important cardiac or respiratory disease
* Any concomitant serious physical illness other than cancer (e.g., immune deficiency disease, bleeding disorder, etc.) within 1 year prior to dosing. No history of autoimmune disease.
* Active, uncontrolled infections within 7 days of study entry requiring systemic therapy.
* Evidence of progression of central nervous system (CNS) metastases or symptomatic CNS metastases within 30 days prior to dosing.
* History of known or suspected autoimmune disease with the specific exceptions of vitiligo, atopic dermatitis, or psoriasis not requiring systemic treatment. (Parts C, D and E only).
* Clinically-significant gastrointestinal disorders, such as perforation, gastrointestinal bleeding, or diverticulitis (Parts D and E only).
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment (Parts D and E only).
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis (Parts D and E only).
* History of interstitial lung disease (Parts D and E only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Adverse events | through 30 days post last dose
  Any adverse change in health or side effect from the initiation of the study drug dose TRX518 monotherapy and TRX518 in combination with gemcitabine, pembrolizumab or nivolumab through completion or premature withdrawal

SECONDARY OUTCOMES:
TRX518 peak concentration (Cmax) | various timepoints through 1 week post dose
  Observations of the distribution, duration of effects and chemical changes of TRX518 monotherapy and TRX518 in combination with gemcitabine, pembrolizumab or nivolumab in the body and the effects and routes of the body's elimination of TRX518
Time to peak concentration (Tmax) | various timepoints through 1 week post dose
  Observations of the distribution, duration of effects and chemical changes of TRX518 monotherapy and TRX518 in combination with gemcitabine, pembrolizumab or nivolumab in the body and the effects and routes of the body's elimination of TRX518
Area under the curve (AUC) | various timepoints through 1 week post dose
  Observations of the distribution, duration of effects and chemical changes of TRX518 monotherapy and TRX518 in combination with gemcitabine, pembrolizumab or nivolumab in the body and the effects and routes of the body's elimination of TRX518
RECIST assessment for evidence of antitumor activity | up to 1 year
  RECIST assessment to determine effects of TRX518 monotherapy and TRX518 in combination with gemcitabine, pembrolizumab or nivolumab on solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Cyndi Sirard, MD, Study Chair — Leap Therapeutics, Inc.
Locations (6):
- United States (6):
  - University of Chicago, Chicago, Illinois
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zappasodi R, Sirard C, Li Y, Budhu S, Abu-Akeel M, Liu C, Yang X, Zhong H, Newman W, Qi J, Wong P, Schaer D, Koon H, Velcheti V, Hellmann MD, Postow MA, Callahan MK, Wolchok JD, Merghoub T. Rational design of anti-GITR-based combination immunotherapy. Nat Med. 2019 May;25(5):759-766. doi: 10.1038/s41591-019-0420-8. Epub 2019 Apr 29. PMID 31036879